CLINICAL TRIAL: NCT06642181
Title: Combined Guanfacine and Mindfulness Meditation as an Adjunct to Buprenorphine Maintenance in Opioid Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Suchismita Ray Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2024002125; 1R61DA059906-01A1 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Mindfulness; Guanfacine; Opioid Use Disorder
Keywords: Opioid; MIndfulness; Guanfacine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Combined Group (Experimental): Will receive both Guanfacine pharmacotherapy and MORE intervention
  Interventions: Drug: Guanfacine pharmacotherapy; Behavioral: Mindfulness Oriented Recovery Enhancement (MORE)
- MORE Group (Experimental): Will receive MORE intervention and placebo medication
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement (MORE)
- Guanfacine Group (Experimental): Will receive Guanfacine intervention and Support group control (non-mindfulness) intervention
  Interventions: Drug: Guanfacine pharmacotherapy
- Control Group (No Intervention): Will receive placebo and support group control (non-mindfulness)

INTERVENTIONS:
Drug: Guanfacine pharmacotherapy — It is a pharmacotherapy
  Arms: Combined Group; Guanfacine Group
Behavioral: Mindfulness Oriented Recovery Enhancement (MORE) — It is a mindfulness intervention
  Arms: Combined Group; MORE Group

SUMMARY:
The US is currently going through an opioid crisis, and while Medication Assisted Treatments such as buprenorphine (BUP) have proved highly effective at stabilizing the neurobiology underlying acute withdrawal, they have been less effective at preventing longer-term relapse and adherence. This may be due to the fact that they do not fully engage the neural processes sub-serving the emotional control of sensitized negative mood and reward sensitivity during stress- and opioid-cue provocation, respectively. In contrast while the alpha2 agonist, guanfacine, may attenuate stress-provoked opioid craving by mediating top-down prefrontal control over sensitized dysphoria, the behavioral intervention, Mindfulness Oriented Recovery Enhancement (MORE) may reduce opioid cue-provoked craving by mediating top-down prefrontal control over hedonic dysregulation. Furthermore, while both interventions separately may prove effective as longer-term adjunctive therapies, they may offer greater efficacy together, providing a unique medication/behavioral combination able to target both stress and reward provocation mechanisms. To optimally test this hypothesis, a staged approach is proposed to first confirm the efficacy of both GXR and MORE, independently and combined (R61), prior to elucidating underlying neural mechanisms (R33). Using a 2 X 2 design, N=80 OUD individuals on BUP will be randomized to either 6-weeks of Guanfacine extended release (GXR; 3mgs, n=40) or placebo (PBO; n=40). Half of all participants in each group will then receive either weekly MORE, or a Support Group (SG) control, creating four intervention groups (Control Grp: PBO+SG, n=20); (GXR Grp: GXR+SG, n=20); (MORE Grp: PBO+ MORE, n=20); (Combined Grp: GXR+MORE, n=20). A pre- and post-laboratory study will be conducted before and after six weeks of intervention where participants will be randomly exposed to 3 personalized guided imageries (stress, opioid cue, neutral). Subjective measures of opioid craving, anxiety, mood, stress, emotional reappraisal, and heart rate will be collected before and after imagery exposure. Following milestone completion, an identical design is proposed in N=144 individuals, where participants will be exposed to imageries in the MRI scanner (R33). On the basis of prior research, it is hypothesized in that GXR will attenuate opioid craving and improve emotion regulation during stress, while MORE will demonstrate the same effects during opioid cue exposure. Combined GXR and MORE will also demonstrate additive or synergistic improvements compared with each intervention alone (R61). The effects of GXR on opioid cue- and MORE on stress-provoked opioid seeking will be explored. In the R33 component, it is hypothesized that GXR will improve regulatory and affective brain function during stress, and MORE will improve regulatory and reward function during opioid cue exposure. Combined GXR and MORE may improve regulatory function in an additive or synergistic manner (R33). Findings will help elucidate the efficacy and neural mechanisms underpinning a novel integrated pharmaco-behavioral therapy for OUD individuals maintained on BUP.

ELIGIBILITY:
Inclusion Criteria:

N=224 individuals with a history of SCID-5 OUD, and maintained on BUP for at least 4 weeks (N=80 in the R61 phase and N=144 in the R33 phase). These individuals must be:

* aged 18 to 55 years and have a body mass index (BMI) of 18-35;
* have a positive urine toxicology screen for non-prescription opioids
* be in good health as verified by screening examination
* able to read English and provide informed consent.

Exclusion Criteria:

* Current SCID V criteria for a moderate to severe substance use disorder other than opioids or nicotine (although mild use will be permitted)
* Use of medications in the last 6 months that may affect cerebral function with the exception of BUP and individuals stabilized on SSRIs
* psychotic or severely psychiatrically disabled (i.e. suicidal, current mania)
* hypotensive individuals with sitting blood pressure below 100/50 mmHG
* Women who are pregnant, nursing or refuse to use a reliable form of birth control
* EKG evidence at baseline screening of any clinically significant conduction abnormalities (Bazett's QTc of >450 msec for men and QTc>470 msec for women)
* R33 phase will additionally include failure to satisfy fMRI safety protocols.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Craving | At pre- and post-intervention (6 weeks intervention)
  Self report of opioid craving will be collected. Will be measured using a likert scale 0 (not at all) to 10 (extreme).
Anxiety | At pre- and post-intervention (6 weeks intervention)
  Self report of anxiety will be collected. Will be measured using a likert scale 0 (not at all) to 10 (extreme). .
Stress | At pre- and post-intervention (6 weeks intervention)
  Self report of stress will be collected. Will be measured using a likert scale 0 (not at all) to 10 (extreme).
Mood | At pre- and post-intervention (6 weeks intervention)
  Self report of mood will be collected. Positive and negative mood will be collected on a 4 point likert scale 0 (not at all) and 4 (extreme)
Emotional Dysregulation | At pre- and post-intervention (6 weeks intervention)
  Self report of emotional dysregulation data will be collected. Will be measured using a 10 point likert scale (0=not at all) and 10 (extreme)
Heart Rate | At pre- and post-intervention (6 weeks intervention)
  Heart rate data will be collected using an EKG monitor during the entire lab procedure while the participants will hear stress, opioid, and neutral related scripts.
Brain Activation | At pre- and post-intervention (6 weeks intervention)
  Brain activation data will be collected using Blood Oxygen Level Dependent (BOLD) signal during functional magnetic resonance imaging (fMRI) while participants hear stress, opioid and neutral scripts.
Brain Connectivity | At pre- and post-intervention (6 weeks intervention)
  Brain connectivity data will be collected using Blood Oxygen Level Dependent (BOLD) signal during functional magnetic resonance imaging (fMRI) while participants hear stress, opioid and neutral scripts.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers School of Health Professions, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT06642181/ICF_000.pdf